CLINICAL TRIAL: NCT04312932
Title: Fatty Acid Supplements Alter Biological Signatures and Behavior in Children With Autism Spectrum Disorder (ASD)
Brief Title: Fatty Acid Supplementation in Children With ASD (Study 2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarah Keim (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Sarah Keim, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB17-00517-2; R33AT009632 (NIH)
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Long chain polyunsaturated fatty acid (LCPUFA) Oil Supplement (Experimental): 25 mg/kg, 50 mg/kg, or 75 mg/kg of gamma-linoleic acid (GLA) + eicosapentaenoic acid (EPA) + docosahexaenoic acid (DHA) as Omega 3-6 oil to be administered twice per day by mouth for 90 days
  Interventions: Drug: LCPUFA Oil Supplement
- Canola Oil (Placebo Comparator): Equal volume (25 mg/kg, 50 mg/kg, or 75 mg/kg) of placebo (canola) oil to be administered twice per day by mouth for 90 days
  Interventions: Dietary Supplement: Canola Oil Placebo

INTERVENTIONS:
Drug: LCPUFA Oil Supplement — 25 mg/kg, 50 mg/kg, or 75 mg/kg of GLA+EPA+DHA as Omega 3-6 oil to be administered twice per day by mouth for 90 days
  Arms: Long chain polyunsaturated fatty acid (LCPUFA) Oil Supplement
Dietary Supplement: Canola Oil Placebo — Equal volume (25 mg/kg, 50 mg/kg, or 75 mg/kg) of placebo (canola) oil to be administered twice per day by mouth for 90 days
  Arms: Canola Oil

SUMMARY:
The objective of the protocol is to test the impact of Omega 3-6 on pre-specified biological signatures (IL-1β, IL-2, and IFNγ) and to correlate changes in the biological signatures with changes in ASD symptoms.

DETAILED DESCRIPTION:
Children with ASD suffer from both mental and physical symptoms that affect quality of life and severely disrupt family well-being. The objective of the protocol is to test the impact of Omega 3-6 on pre-specified biological signatures (IL-1β, IL-2, and IFNγ) and to correlate changes in the biological signatures with changes in ASD symptoms. Fatty acid supplements are natural products with anti-inflammatory properties often used for treatment of ASD symptoms, but the efficacy remains unproven.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-6 years old
* ASD diagnosis at Nationwide Children's Hospital within the prior 6 months
* English is primary language

Exclusion Criteria:

* Fatty acid supplementation in the past 6 months
* Consumes fatty fish more than 3 times per week
* Still breastfeeding or formula feeding
* Bleeding disorder
* Quadriparesis
* Deafness
* Blindness
* Seizure disorder diagnosis
* Autoimmune disorder including Type 1 Diabetes, Fragile X, Rett, Angelman Syndromes, Tuberous Sclerosis
* Feeding problems precluding consumption of the supplement
* Ingredient allergy (canola, fish, or borage seed)
* Planned surgeries scheduled within the time frame of trial participation

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Keim, PhD, Principal Investigator — Nationwide Children's Hospital; Lynette Rogers, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- GLA + EPA + DHA Group: 50 mg/kg of gamma-linoleic acid (GLA) + eicosapentaenoic acid (EPA) + docosahexaenoic acid (DHA) as Omega 3-6 oil to be administered twice per day by mouth for 90 days
  LCPUFA Oil Supplement: 50 mg/kg of GLA+EPA+DHA as Omega 3-6 oil to be administered twice per day by mouth for 90 days
- Canola Oil Group: Assignment an equivalent volume of canola oil as the GLA+EPA+DHA group, based on body weight.
Period: Overall Study
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Started | 48 | 50
Completed | 45 | 46
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48 | 48 | 96
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 37 | 37 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 45 | 44 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 9 | 20
  White | 28 | 28 | 56
  More than one race | 5 | 9 | 14
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Pervasive Developmental Disorder Behavior Inventory (PDDBI) - Autism Composite
Description: Change in PDDBI Autism Composite raw score. This scale measures the severity and nature of autism symptoms. Autism Composite raw scores range -31 to 262. Higher scores indicate greater severity. We omitted the Semantic/Pragmatic Problems subscale from the calculation of the PDD autism composite raw score because including that subscale penalizes children who are nonverbal at baseline but gain language during the study.
Time Frame: Baseline to 90 days post randomization.
Measure: Mean (Standard Deviation); unit: raw score on a scale
Arm/Group | Long Chain Polyunsaturated Fatty Acid (LCPUFA) Oil Supplement | Canola Oil
Number analyzed (Participants) | 48 | 48
raw score on a scale
  Baseline | 115.5 (32.5) | 106.5 (34.6)
  90 days post randomization (End of Trial) | 98.1 (34.1) | 91.4 (36.1)

2. Secondary Outcome: Vineland Adaptive Behavior Scales 2nd ed. (Modified Timeframe of 90 Days) Adaptive Behavior Composite
Description: Change in adaptive behavior composite score. These are raw scores. Each one is a sum of its component subdomain raw scores. Lower scores indicate lower adaptive level. Scores range 0-634.
Time Frame: Baseline to 90 days post randomization (End of Trial)
Measure: Mean (Standard Deviation); unit: raw score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 48 | 48
raw score on a scale
  Baseline | 280.3 (99.89) | 277.1 (114.8)
  90 days post randomization (End of Trial) | 303.6 (116.9) | 290.0 (120.3)

3. Secondary Outcome: Pervasive Developmental Disorder (PDD) Behavior Inventory (PDDBI) - Aggressiveness Problems
Description: Change in PDDBI Aggressiveness Problems raw score. Aggressiveness domain looks at self-directed aggressive behaviors, incongruous negative affect, problems when caregiver returns from an outing, aggressiveness towards others, and overall temperament problems. Aggressiveness raw scores range from 0-60; higher scores are indicative of more aggressiveness.
Time Frame: Baseline to 90 days post randomization.
Measure: Mean (Standard Deviation); unit: raw score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 48 | 48
raw score on a scale
  Baseline | 26.7 (13.2) | 26.5 (13.8)
  90 days post randomization (End of Trial) | 23.1 (12.6) | 23.8 (13.4)

4. Secondary Outcome: Preschool Language Scales - 5 (PLS-5) Auditory Comprehension
Description: Changes in Auditory Comprehension raw score. Higher scores represent better child comprehension of language. Raw scores range 0-65 for Auditory Comprehension.
Time Frame: Baseline to 90 days post randomization.
Measure: Mean (Standard Deviation); unit: raw score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 48 | 48
raw score on a scale
  Baseline | 29.4 (14.3) | 28.9 (13.6)
  90 days post randomization (End of Trial) | 30.3 (14.9) | 30.3 (13.8)

5. Secondary Outcome: Childhood Autism Rating Scale (CARS2) (2nd ed.)
Description: Changes in Continuous Total (raw) Score. (higher scores indicate greater symptoms) Range 15-60.
Time Frame: Baseline to 90 days post randomization.
Measure: Mean (Standard Deviation); unit: raw score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 48 | 48
raw score on a scale
  Baseline | 32.9 (8.1) | 30.9 (7.5)
  90 days post randomization (End of Trial) | 32.4 (7.5) | 31.5 (7.8)

6. Secondary Outcome: Autism Impact Measure - Total
Description: The Autism Impact Measure is a newly developed instrument for measuring change in Autism Spectrum Disorder related behaviors. (Houghton, Journal of Autism and Developmental Disorders, 2019). The Autism Impact Measure (AIM) Total Score represents the overall level of autism symptom impact across all measured domains, incorporating both the frequency and impact of symptoms. The possible range of raw scores for the AIM Total is 41 to 410. This scale measures the global severity and pervasiveness of autism-related behaviors, with higher scores indicating greater symptom impact and worse functioning, and lower scores reflecting fewer symptoms and better functioning.
Time Frame: Baseline to 90 days post randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 45 | 43
score on a scale
  Baseline | 222.4 (45.5) | 215.6 (55.5)
  90 days post randomization (End of Trial) | 207.9 (50.6) | 200.0 (55.7)

7. Secondary Outcome: Preschool Language Scales-5 Expressive Communication
Description: Changes in Expressive Communication raw score. Higher scores represent better child ability to communicate with others. Raw scores range 0-67.
Time Frame: Baseline (day 0) to end of trial (90 days)
Measure: Mean (Standard Deviation); unit: raw score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 48 | 48
raw score on a scale
  baseline day 0 | 31.0 (11.5) | 28.8 (10.5)
  end of trial day 90 | 31.2 (12.2) | 30.7 (11.9)

8. Secondary Outcome: Preschool Language Scales-5 Total Language
Description: Changes in Total Language raw score (sum of Auditory Comprehension and Expressive Communication raw scores). Higher scores represent better communication ability. Raw scores range 0-131.
Time Frame: Baseline (day 0) to end of trial (90 days)
Measure: Mean (Standard Deviation); unit: raw score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 48 | 48
raw score on a scale
  baseline day 0 | 60.4 (25.3) | 57.6 (23.2)
  end of trial day 90 | 61.5 (26.6) | 61.0 (25.2)

9. Secondary Outcome: Autism Impact Measure - Restricted Behavior
Description: The Autism Impact Measure (AIM) Repetitive Behavior Score assesses repetitive movements, rituals, and restricted interests, capturing both how often these behaviors occur and how much they affect daily life. The possible range of raw scores for this scale is 16 to 80. It measures the frequency and impact of repetitive behaviors, with higher scores reflecting more frequent and disruptive behaviors and poorer functioning.
Time Frame: Baseline to 90 days post randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 45 | 43
score on a scale
  Baseline | 43.3 (11.3) | 43 (14.3)
  90 days post randomization (End of Trial) | 40.3 (12.4) | 38.3 (12.3)

10. Secondary Outcome: Autism Impact Measure - Communication
Description: The Autism Impact Measure (AIM) Communication Score evaluates expressive and receptive communication skills, taking into account both the frequency of communication challenges and their impact on functioning. The possible range of raw scores for this scale is 12 to 60. It measures how effectively an individual communicates, with higher scores indicating greater communication difficulties and worse functioning.
Time Frame: Baseline to 90 days post randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 45 | 43
score on a scale
  Baseline | 36.4 (11.1) | 37.1 (10.1)
  90 days post randomization (End of Trial) | 32.9 (11.4) | 35.4 (10.4)

11. Secondary Outcome: Autism Impact Measure - Atypical Behavior
Description: The Autism Impact Measure (AIM) Atypical Behavior Score captures unusual sensory responses, emotional regulation difficulties, and other atypical behaviors, assessing both how often these behaviors occur and how much they interfere with daily life. The possible range of raw scores for this scale is 12 to 60. It measures the presence and impact of atypical behaviors, with higher scores indicating more frequent or intense atypical behaviors and poorer functioning.
Time Frame: Baseline to 90 days post randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 45 | 43
score on a scale
  Baseline | 30.2 (9.6) | 29.5 (9.4)
  90 days post randomization (End of Trial) | 28.7 (9.5) | 26 (9.5)

12. Secondary Outcome: Autism Impact Measure - Social Reciprocity
Description: The Autism Impact Measure (AIM) Social Reciprocity Score assesses social engagement, emotional responsiveness, and reciprocal interactions, considering both the frequency and impact of social difficulties. The possible range of raw scores for this scale is 10 to 50. It measures social responsiveness and connectedness, with higher scores indicating greater social difficulty and worse functioning.
Time Frame: Baseline to 90 days post randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 45 | 43
score on a scale
  Baseline | 26.8 (6.2) | 25.5 (7.9)
  90 days post randomization (End of Trial) | 25.4 (7) | 24.3 (8.4)

13. Secondary Outcome: Autism Impact Measure - Peer Interaction
Description: The Autism Impact Measure (AIM) Peer Interaction Score evaluates social interest, initiation, and quality of interactions with peers, capturing both how often behaviors occur and how impactful they are. The possible range of raw scores for this scale is 8 to 40. It measures the child's ability to interact appropriately with peers, with higher scores indicating more challenges in peer relationships and worse functioning. for this scale is 10 to 50. Higher scores indicating greater social difficulty and worse functioning.
Time Frame: Baseline to 90 days post randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 45 | 43
score on a scale
  Baseline | 26.8 (6.2) | 25.5 (7.9)
  90 days post randomization (End of Trial) | 25.4 (7) | 24.3 (8.4)

14. Secondary Outcome: Vineland Adaptive Behavior Scales 2nd ed. (Modified Timeframe of 90 Days) Communication
Description: Change in communication score. These are raw scores. Each one is a sum of its component subdomain raw scores. Lower scores indicate lower adaptive level. Scores range 0-148.
Time Frame: Baseline to 90 days post randomization (End of Trial)
Measure: Mean (Standard Deviation); unit: raw score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 45 | 43
raw score on a scale
  Baseline | 74.2 (39.4) | 67.9 (39.6)
  90 days post randomization (End of Trial) | 80 (42.6) | 73.4 (39.4)

15. Secondary Outcome: Vineland Adaptive Behavior Scales 2nd ed. (Modified Timeframe of 90 Days) Socialization
Description: Change in socialization score. These are raw scores. Each one is a sum of its component subdomain raw scores. Lower scores indicate lower adaptive level. Scores range 0-174.
Time Frame: Baseline to 90 days post randomization (End of Trial)
Measure: Mean (Standard Deviation); unit: raw score on a scale
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
Number analyzed (Participants) | 45 | 43
raw score on a scale
  Baseline | 64.4 (30) | 66.1 (34.8)
  90 days post randomization (End of Trial) | 67.9 (31.8) | 68.5 (35.8)

ADVERSE EVENTS:
Time Frame: 90 days
Description: Safety Monitoring Uniform Report Form (SMURF)
Arm/Group | GLA + EPA + DHA Group | Canola Oil Group
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 45/48 | 46/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLA + EPA + DHA Group (N=48) | Canola Oil Group (N=48)
Chest or breathing (Respiratory, thoracic and mediastinal disorders) | 25 (42) | 25 (41)
Ears (Ear and labyrinth disorders) | 8 (8) | 4 (5)
Energy level (Metabolism and nutrition disorders) | 10 (10) | 6 (6)
Eyes (Eye disorders) | 0 (0) | 1 (1)
Genitourinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Gastrointestinal and eating (Gastrointestinal disorders) | 36 (63) | 37 (77)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Heart (Cardiac disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 14 (18) | 14 (15)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Mouth lips teeth (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal and movement (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Nose, sinus, throat (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 13 (15)
Psychological (Psychiatric disorders) | 29 (46) | 26 (47)
Skin or hair (Skin and subcutaneous tissue disorders) | 8 (10) | 9 (11)
Sleep (Psychiatric disorders) | 19 (20) | 11 (12)

LIMITATIONS AND CAVEATS:
This trial may have been underpowered to detect a clinically meaningful effect on autism symptoms. 90 days is short and this may have precluded observing effects. The focus on children with confirmed autism diagnoses and English language limit the generalizability to older or non-English speaking children or those with subclinical autistic traits. The single site-specific context may not be representative of other settings. Compliance with consuming the daily supplement was challenging.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT04312932/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT04312932/ICF_001.pdf